CLINICAL TRIAL: NCT04651062
Title: Detection of Adenomas in Screening Colonoscopy - Endocuff Study
Brief Title: Detection of Adenomas in Screening Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herning Hospital (Other)
Responsible Party: Principal Investigator, Claudia Jaensch, principan investigator, Herning Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-16-02-828-17
Record Dates: First submitted 2018-03-01; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Adenoma Colon
Keywords: adenoma detection rate; screening colonoscopy

STUDY DESIGN:
Intervention Model Description: this is a randomized controlled trial
Masking Description: participant, care provider, investigator and outcomes assessor know whether or not a endocuff has been used for the colonoscopy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endocuff (Experimental): all patients having performed a screeningscolonoscopy and being randomized to colonoscopy with the use of endocuff
  Interventions: Device: endocuff
- no cuff (Active Comparator): all patients participating in a screeningscolonoscopy being randomized to colonoscopy without the use of endocuff
  Interventions: Procedure: no endocuff

INTERVENTIONS:
Device: endocuff — Endocuff is a relatively new device which is intended to be attached to the end of the colonoscope.
  Arms: endocuff
Procedure: no endocuff — colonoscopy is performed without endocuff.
  Arms: no cuff

SUMMARY:
The Endocuff study aims to show an increase of the number of detected adenomas in screening colonoscopies when a endocuff vision (Arc Medical Design Ldt Leeds England) is used.

DETAILED DESCRIPTION:
Endocuff is a relatively new device which is intended to be attached to the end of the colonoscope. Several minor studies have shown that the use of Endocuff probably increases the number of detected polyps in colonoscopy. Endocuff is made of soft plastic and has been designed to give an optimal view of the entire colon. It gently averts and flattens folds in order to see small polyps "hiding" in the space behind colonic folds.

The purpose of this study is to investigate into the effect of the Endocuff in screening colonoscopy compared with screening colonoscopy performed without Endocuff. The device has been used during several years yet an effect on the number of polyps detected during screenings colonoscopy has not been shown. This studies main hypothesis is that the use of Endocuff in screenings colonoscopy will increase the adenoma detection rate in these patients, with a potential to reduce interval cancer.

This study is a randomized controlled trial with 900 patients.

ELIGIBILITY:
Inclusion Criteria:

* all Citizens participating in the national bowel screening program

Exclusion Criteria:

* persons who are disabled and who do not understand the Danish language
* persons treated with Marcoumar, Marevan, Eliquis, Pradaxa e.g. and who are not eligible to polyp resection
* persons who due to diseases of the eyes or Heart are not allowed to receive Buscopan.
* persons with active colitis/diverticulitis, colon stenosis e.g. due to cancer, where a complete colonoscopy is not possible to achieve

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1178 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
adenoma | 2 weeks
  number of adenomas found during colonoscopy

SECONDARY OUTCOMES:
cecal intubation rate | up to 2 hours
  is the cecum reached during the colonoscopy
cecal intubation time | up to 2 hours
  number of minutes from start procedure to cecum reached
withdrawal time | up to 60 minutes
  number of minutes from cecum reached to end of the procedure, only if no polyps are found
adenoma size | up to 4 weeks
  size of adenomas detected
adenoma site | up to 4 weeks
  where in the bowel the adenoma was detected

CONTACTS AND LOCATIONS:
Locations (1):
- Kirurgisk Afdeling, Herning, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jaensch C, Jepsen MH, Christiansen DH, Madsen AH, Madsen MR. Adenoma and serrated lesion detection with distal attachment in screening colonoscopy: a randomized controlled trial. Surg Endosc. 2022 Sep;36(9):1-9. doi: 10.1007/s00464-022-09049-5. Epub 2022 Feb 9. PMID 35141776